CLINICAL TRIAL: NCT02954588
Title: The Effect of Pyridoxamine Supplementation on Vascular Function and Insulin Sensitivity; a Double-blind Randomized Placebo Controlled Trial in Abdominally Obese Subjects.
Brief Title: Effect of Pyridoxamine Supplementation on Vascular Function and Insulin Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Top Institute Food and Nutrition (Other); Center for Translational Molecular Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: NL51023.068.16
Record Dates: First submitted 2016-11-02; First posted 2016-11-03 (Estimated); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Abdominal Obesity Metabolic Syndrome
MeSH Terms: conditions — Abdominal obesity metabolic syndrome | interventions — Pyridoxamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Pyridoxamine (1) (Active Comparator): Subjects will be asked to consume dietary supplements containing pyridoxamine (dosage 1), three times daily during 8 weeks.
  Interventions: Dietary Supplement: Pyridoxamine
- Pyridoxamine (2) (Active Comparator): Subjects will be asked to consume dietary supplements containing pyridoxamine (dosage 2), three times daily during 8 weeks
  Interventions: Dietary Supplement: Pyridoxamine
- Placebo (Placebo Comparator): Subjects will be asked to consume dietary supplements containing placebo (amylum solani), three times daily during 8 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Pyridoxamine
  Arms: Pyridoxamine (1); Pyridoxamine (2)
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
A growing body of evidence demonstrates that increased adipose mass, especially visceral adipose tissue, contributes directly towards an increase in systemic inflammation, (micro-)vascular dysfunction and the burden of cardiovascular disease (CVD), insulin resistance and type 2 diabetes. Advanced glycation/lipoxidation endproducts (AGEs/ALEs) are a heterogeneous family of unavoidable by-products, which are formed by reactive metabolic intermediates derived from glucose and lipid oxidation. In addition to the overwhelming amount of data demonstrating the role of AGEs/ALEs in the development of (micro-)vascular dysfunction and disease, accumulation of AGEs/ALEs in the expanding adipose tissue contributes to the dysregulation of adipokines and the development of insulin resistance.

The investigators want to examine, in a double-blind randomized placebo controlled parallel study, the physiological effect of a dietary intervention with pyridoxamine in abdominally obese persons.

A sub-study is implemented next to the clinical trial. The objective of the sub-study is to measure the metabolization and kinetics of pyridoxamine in plasma and urine with UPLC-MS/MS. The sub-study comprises of 5 additional healthy volunteers, with pyridoxamine as an oral supplement.

ELIGIBILITY:
Inclusion Criteria:

* Abdominal obesity: Waist circumference for men should be above 102 cm and for women above 88 cm.
* Caucasian (because of skin fluorescence and capillary microscopy measurements)
* Aged 18-75 years

Exclusion Criteria:

* Diabetes (i.e. using anti-diabetic medication, fasting glucose >7.0 mmol/L, HbA1c >6.5%).
* Active or history of cardiovascular disease (e.g. stroke, coronary artery disease, peripheral vascular disease, congestive heart failure, cardiac shunts, cardiac surgery, pulmonary hypertension, cardiac arrhythmias, family history of cardiac arrhythmias or sudden cardiac death)
* Hyperlipidemia (defined as serum total cholesterol > 8 mmol/L or TG > 4 mmol/L)
* Smoking (>10 cigarettes per day)
* High alcohol usage (>4 U/day) or drug abuse
* Use of medication known to influence glucose metabolism, vascular function (e.g. glucocorticosteroids, NSAID's)
* Higher grade hypertension (> 179 mmHg SBP and/or > 109 mmHg DBP) in order not to expose subjects to unnecessary risks)
* Known allergic reaction to ultrasound contrast-agent
* Pulmonary or inflammatory disease
* Kidney failure or electrolyte disorders
* Use of dietary supplements or an investigational product within the previous month
* Unstable body weight (no drastic changes in life style before or during the intervention are allowed, this means no weight gain or loss >3 kg in the last two months)
* Pregnancy or lactation
* No change in use of oral anticonceptiva or IUD (12 weeks prior of during the intervention)
* Unwillingness to give up being a blood donor (or having donated blood) from 8 weeks prior to the start of the study and during the study
* Insufficient knowledge of the Dutch language

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2016-10-14 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-08-08 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | Difference after 8 weeks of intervention
  Assessed by hyperinsulinemic-euglycemic clamp
Microvascular function | Difference after 8 weeks of intervention
  Assessed by contrast-enhanced ultrasound (CEUS) in skeletal muscle

CONTACTS AND LOCATIONS:
Overall Officials: Casper G Schalkwijk, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands

REFERENCES:
- [Derived] Van den Eynde MDG, Scheijen JLJM, Stehouwer CDA, Miyata T, Schalkwijk CG. Quantification of the B6 vitamers in human plasma and urine in a study with pyridoxamine as an oral supplement; pyridoxamine as an alternative for pyridoxine. Clin Nutr. 2021 Jul;40(7):4624-4632. doi: 10.1016/j.clnu.2021.05.028. Epub 2021 Jun 10. PMID 34229268